CLINICAL TRIAL: NCT01088347
Title: A Phase 1b/2 Study With the Agonistic TRAIL-R1 Antibody, Mapatumumab, in Combination With Cisplatin and Radiotherapy as a First Line Therapy in Patients With Advanced Cervical Cancer.
Brief Title: Mapatumumab, Cisplatin and Radiotherapy for Advanced Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-11-2009 (versions 2.0); 2009-015941-22 (EudraCT Number)
Record Dates: First submitted 2010-03-10; First posted 2010-03-17 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Cervical Cancer
Keywords: TRAIL; TRM1; advanced cervical cancer; mapatumumab; Uterine cervical neoplasm; Radiotherapy; Cisplatin
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — mapatumumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Advanced cervical cancer patients (Experimental)
  Interventions: Drug: mapatumumab; Drug: cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: mapatumumab — Mapatumumab (10 or 30 mg/kg) intravenously on days 1, 22, and 45. In phase 2 the MTD established in phase 1 will be used.
Drug: cisplatin — Cisplatin 40 mg/m2 intravenously on days 8, 15, 22, 29, 36, and 45
Radiation: radiotherapy — Radiotherapy: a total dose of 45 Gy will be given in fractions of 1.8 Gy, five fractions per week (days 8-12, 15-19, 22-26, 29-33, and 36-40), by external beam irradiation by photon beam of at least 6 MV. After completing the five weeks of external beam irradiation, evaluation will take place to determine whether the boost can be given by brachytherapy. If brachytherapy is not feasible, the boost will be given by external beam irradiation to a total dose of 70.2 Gy in fractions of 1.8 Gy.

SUMMARY:
Chemoradiotherapy has become the standard of care for women with locally advanced cervical cancer. The available data support a 30 to 50% reduction in the risk of death from cervical cancer for women with locally advanced disease undergoing radiotherapy (RT) and concomitant cisplatin-based chemotherapy compared to RT alone. Despite the fact that this is currently the best treatment of locally advanced cervical cancer, 5-year overall survival is still only 52%.

The fully human, agonist monoclonal antibody mapatumumab binds to the Tumor necrosis factor-Related Apoptosis-Inducing Ligand Receptor 1 (TRAIL-R1, DR4) and induces cytotoxicity in multiple tumor cell lines in vitro and in vivo. In multiple phase I and phase II studies, mapatumumab appeared to be safe both as single agent and in combination with chemotherapy, including cisplatin.

In cervical cancer cell lines, mapatumumab induced apoptosis in 51% of the cells. Mapatumumab in combination with irradiation increased apoptosis to 83%.

In this phase 1b/2 study, the investigators will evaluate the safety, tolerability and efficacy of mapatumumab in combination with cisplatin and radiotherapy in patients with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed stage IB2, IIA2, IIB, III, and IVA cervical cancer, according to the FIGO classification
2. Adequate bone marrow, renal and liver function:

   * Absolute neutrophil count ≥ 1.5 x 109 /L.
   * Platelet count ≥ 100 x 109 /L.
   * Serum creatinine level ≤ 1.5 x upper limit of normal (ULN).
   * Total bilirubin < 1.25 x ULN.
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN.
3. Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
4. Age 18 years or older.
5. Life expectancy of ≥ 12 weeks.
6. Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the study and follow-up procedures.

Exclusion Criteria:

1. Any co-morbid condition that in the judgment of the investigator renders the subject at high risk of treatment complications or reduces the possibility of assessing clinical effect.
2. Cytotoxic agent, hormonal therapy, or radiation therapy within 3 weeks (6 weeks for nitrosoureas or mitomycin-C) prior to day 1, cycle 1; investigational agent within 4 weeks prior to day 1, cycle 1.
3. Need for concomitant anticancer therapy (surgery, radiation therapy, chemotherapy, immunotherapy, radiofrequency ablation) or other investigational agents during the study treatment period.
4. Major surgery within 4 weeks before enrollment; minor surgery (except for insertion of vascular access device) within 2 weeks before enrollment; or not yet recovered from the effects of the surgery.
5. Systemic steroids within 1 week before enrollment except steroids used as part of an antiemetic regimen or maintenance-dose steroids for non-cancerous disease.
6. History of any infection requiring hospitalization or antibiotics within 2 weeks before enrollment.
7. Known brain or spinal cord metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and steroids.
8. Known human immunodeficiency virus infection.
9. Unstable angina, myocardial infarction, cerebrovascular accident, > Class II congestive heart failure according to the New York Heart Association Classification for Congestive Heart Failure within 6 months before enrollment.
10. Pregnant female or nursing mother.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Phase 1b: safety and tolerability of mapatumumab in combination with cisplatin and radiotherapy Phase 2: efficacy of mapatumumab in combination with cisplatin and radiotherapy | 5 months
  Phase 2: pathological complete response rate

SECONDARY OUTCOMES:
Disease free survival, overall survival | From enrollment until recurrence of disease, from enrollment until death
Apoptotic pathway biomarkers, PK parameters | During the study, until 5 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD,PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Maduro JH, de Vries EG, Meersma GJ, Hougardy BM, van der Zee AG, de Jong S. Targeting pro-apoptotic trail receptors sensitizes HeLa cervical cancer cells to irradiation-induced apoptosis. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):543-52. doi: 10.1016/j.ijrobp.2008.06.1902. PMID 18793956
- [Background] Mom CH, Verweij J, Oldenhuis CN, Gietema JA, Fox NL, Miceli R, Eskens FA, Loos WJ, de Vries EG, Sleijfer S. Mapatumumab, a fully human agonistic monoclonal antibody that targets TRAIL-R1, in combination with gemcitabine and cisplatin: a phase I study. Clin Cancer Res. 2009 Sep 1;15(17):5584-90. doi: 10.1158/1078-0432.CCR-09-0996. Epub 2009 Aug 18. PMID 19690193